CLINICAL TRIAL: NCT02265406
Title: PROPHY-VAP: Prevention of Early Ventilation Acquired Pneumonia (VAP) in Brain Injured Patients by a Single Dose of Ceftriaxone
Acronym: PROPHY-VAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROPHY-VAP
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Early Ventilation Acquired Pneumonia in Brain Injured Patients
MeSH Terms: interventions — Anti-Infective Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ceftriaxone (Experimental)
  Interventions: Drug: Anti-Infective Agents
- Sodium Chloride (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anti-Infective Agents
  Arms: Ceftriaxone
Drug: Placebo
  Arms: Sodium Chloride

SUMMARY:
Ventilation-associated pneumonia (VAP) is the main site of healthcare-associated infections in the brain injured patients, with an incidence rate of 22% to 58%. VAP increases morbi-mortality, length of stay in intensive care and overall management costs. The prevention of ICU nosocomial infections depends on several measures : orotracheal intubation route, maintaining tube cuff pressure between 25 and 30 cm of water (H2O), maintaining a semi-seated position >= 30°, nasal and oropharyngeal care at regular intervals, striving to avoid unscheduled extubation, and use of a written sedation-analgesia algorithm allowing for early weaning from ventilation. Two randomized study show that administration of antibiotic therapy after intubation reduces the risk of early VAP incidence. However, in clinical practice, its administration solely purposes of limiting VAP occurence is not presently recommended. Indeed, to date no placebo blind controlled study was been realized and the fear of development of bacterial resistance remains stronger than the efficiency of this prevention measure. This aim of the present study is to show by a placebo randomized study that 2g of Ceftriaxone within 8 hours post-intubation after a brain injury decrease the risk of occurence an early VAP.

Ancillary study An ancillary study is performed in 2 centres which routinely practice rectal swabs at admission and discharge of ICU, to survey intestinal flora (CHU of Angers and CHU of Rennes). The goal of this study is to compare the incidence of acquired cephalosporin resistant gram negative bacteria at the discharge of ICU between the 2 groups of patients, receiving or not ceftriaxone.

ELIGIBILITY:
Inclusion Criteria:

* Brain injured patients with a Glasgow scale score ≤ 12 who require ventilation more than 48 hours

Exclusion Criteria:

* Patient with a high risk of death within the 48 first hours after admission,
* Patient intubated for more than12 hours
* Intubation after the 48th hours after admission
* Coverage to cardiopulmonary arrest
* Coma due to a tumor, an infectious disease or a cardiac arrest
* Previous hospitalisation within the last month before admission for coma
* béta-lactamines allergy
* Patient who receive already antibiotics at the admission for a previous infection
* Prophylactic antibiotic due to be done within 24 hours following the randomisation
* Patient Intubated through a tracheal tube with subglottic secretion aspiration
* Patient with a tracheotomy
* Patient or family refuse to be involved in the study
* Use of Ceftriaxone within 2 days before enrolment
* Participation in another research protocol focusing on an anti-infective treatment or on a measure decreasing the risk of infection
* Patients not affiliated to a social security scheme, Pregnant woman or breast-feeding mother, Patients deprived of their liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-07-25 (Actual)

PRIMARY OUTCOMES:
Incidence of early VAP, proportion of patients who develop a VAP within the 7 first day after mechanical ventilation (the 7th day included), confirm with microbiological culture, within all included patients. | 30 months

SECONDARY OUTCOMES:
- Incidence of late VAP (> 7 jours) | 30 months
- Global incidence of VAP during intensive care period (limited to day 60) | 30 months
- Type of bacteria and their sensitivity for early or late VAP, | 30 months
- Time between inclusion and occurence of the first VAP (limited to day 28), | 30 months
- Length of the first period of mechanical ventilation during the intensive care period, | 30 months
- Time between inclusion and the first spontaneous ventilation test (limited to day 28), | 30 months
- Length of antibiotherapy during intensive care period, | 30 months
- Length of intensive care, limited to 60 days, | 30 months
- Length of stay in intensive care unit, limited to 60 days, | 30 months
- Length of stay at the hospital, limited to 60 days, | 30 months
- Neurological prognosis at the discharge of the intensive care unit, | 30 months
- Mortality at day 28 and 60. | 30 months
- Incidence of ventilated associated event (limited to day 60) | 30 months
- Comparison of the global incidence of VAP according to the diagnosis defined by "American Thoracic Society" or by "Centers for Disease Control" | 30 months

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - University Hospital of Angers, Angers
  - CHU, Bordeaux
  - CHRU, Montpellier
  - University Hospital of Nantes, Nantes
  - University Hospital of Poitiers, Poitiers
  - University Hospital of Rennes, Rennes
  - Thomas GEERAERTS, Toulouse
  - Djilali ELAROUSSI, Tours

REFERENCES:
- [Derived] Dahyot-Fizelier C, Lasocki S, Kerforne T, Perrigault PF, Geeraerts T, Asehnoune K, Cinotti R, Launey Y, Cottenceau V, Laffon M, Gaillard T, Boisson M, Aleyrat C, Frasca D, Mimoz O; PROPHY-VAP Study Group and the ATLANREA Study Group. Ceftriaxone to prevent early ventilator-associated pneumonia in patients with acute brain injury: a multicentre, randomised, double-blind, placebo-controlled, assessor-masked superiority trial. Lancet Respir Med. 2024 May;12(5):375-385. doi: 10.1016/S2213-2600(23)00471-X. Epub 2024 Jan 20. PMID 38262428
- [Derived] Dahyot-Fizelier C, Frasca D, Lasocki S, Asehnoune K, Balayn D, Guerin AL, Perrigault PF, Geeraerts T, Seguin P, Rozec B, Elaroussi D, Cottenceau V, Guyonnaud C, Mimoz O; PROPHY-VAP Study group, ATLANREA group. Prevention of early ventilation-acquired pneumonia (VAP) in comatose brain-injured patients by a single dose of ceftriaxone: PROPHY-VAP study protocol, a multicentre, randomised, double-blind, placebo-controlled trial. BMJ Open. 2018 Oct 18;8(10):e021488. doi: 10.1136/bmjopen-2018-021488. PMID 30341115